CLINICAL TRIAL: NCT01575184
Title: Effect of Shoulder Position and Head Rotation on Size and Relative Position of Internal Jugular Vein to Carotid Artery in Infants and Children
Brief Title: Effect of Shoulder Traction on Size and Relative Position of Internal Jugular Vein to Carotid Artery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Assistant Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SMC 2011-04-004-001
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Internal Jugular Vein Cannulation; Common Carotid Artery; Infants
Keywords: internal jugular vein cannulation; common carotid artery; infants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shoulder traction (Experimental): The ultrasonographic measurements with shoulder traction
  Interventions: Other: caudo-ipsilateral traction of shoulder
- No traction (Active Comparator): The ultrasonographic measurements without shoulder traction
  Interventions: Other: The ultrasonographic measurements without shoulder traction

INTERVENTIONS:
Other: caudo-ipsilateral traction of shoulder — After the head rotation (0, 40, 80 degrees) to the contralateral side from the ultrasound measuring site, the slight caudo-ipsilateral traction of shoulder will be applied without changing the degree of the head rotation.
  Arms: Shoulder traction
Other: The ultrasonographic measurements without shoulder traction — After the head rotation (0, 40, 80 degrees) to the contralateral side from the ultrasound measuring site, the no traction of shoulder will be applied.
  Arms: No traction

SUMMARY:
Internal jugular vein (IJV) catheterization is frequently performed in infants undergoing major surgery. Although it has been suggested that head rotation increases the degree of overlapping between IJV and carotid artery (CA), IJV catheterization without head rotation is extremely difficult in infants. The aim of the present study is to evaluate whether the caudo-lateral traction of the ipsilateral arm can decrease the degree of overlapping between IJV and CA in infants during head rotation.

DETAILED DESCRIPTION:
Central venous catheterization is frequently performed in pediatric patients undergoing major surgery for fluid management and vasoactive drug therapy. Compared to subclavian vein, internal jugular vein (IJV) is generally preferred for catheterization because of the low incidence of serious complications, such as pneumothorax and hemothorax. However, especially in infants, IJV catheterization is still technically difficult because of the small size of the vein and anatomical variation.

In previous studies, ultrasound guidance and keeping in neutral head position have been recommended to increase the success rate and to decrease the overlap between carotid artery (CA) and IJV, respectively. However, devices for ultrasonography are not always available. Moreover, IJV catheterization without head rotation could be extremely difficult in infants because of relative the larger skull and the smaller neck than those of adults. Therefore, a simple method to relieve the overlap between CA and IJV would be needed.

During head rotation to the contralateral side, the cephalic part of IJV is moved to the same direction. Accordingly, the investigators thought that the counter traction of the caudal part of IJV using the caudo-lateral traction of the ipsilateral arm might relieve the overlap caused from head rotation. Therefore, the investigators evaluated the effect of the caudo-lateral traction of the ipsilateral arm on the overlap between common CA and IJV in infants.

ELIGIBILITY:
Inclusion Criteria:

* infants undergoing elective surgery

Exclusion Criteria:

* subjects with congenital heart disease or mass in head and neck
* Subjects with anatomical malformation of great vessels
* previous central venous access via IJV

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Carotid artery (CA) overlap (%) | 10 seconds after head positioning
  CA overlap = (overlap distance between CA and internal jugular vein)/CA diameter) × 100 measured by ultrasound image

SECONDARY OUTCOMES:
IJV (internal jugular vein) safety portion (%) | 10 seconds after head positioning
  IJV safety portion = (1-ovelap distance/IJV diameter) × 100 measured by ultrasound image
overlap distance (mm) | 10 seconds after head position
  overlap distance (mm) of carotid artery and internal jugular vein measured by ultrasound image
jugular to carotid distance (mm) | 10 seconds after head position
  the distance (mm) between lateral border of carotid artery and center of internal jugula vein measured by ultrasound image
CA diameter (mm) | 10 seconds after head positioning
  carotid artery diameter (mm) measured by ultrasound image
IJV diameter (mm) | 10 seconds after head positioning
  internal jugualr vein diameter (mm) measured by ultrasound image

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hwan Lee, MD, PhD, Principal Investigator — Samsung Medical Center; Won Ho Kim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea